CLINICAL TRIAL: NCT00593086
Title: The Use of Virtual Reality Video Games to Control Procedural Pain During Burn Wound Care
Brief Title: Virtual Reality in Burn Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-06-024
Record Dates: First submitted 2007-12-26; First posted 2008-01-14 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Burns; Pain
Keywords: wound care
MeSH Terms: conditions — Burns; Pain | interventions — Pain Management; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Standard of care pain management
  Interventions: Procedure: Pain management; Other: Standard of care/no virtual reality game
- B (Experimental): SnoWorld Virtual Reality Game
  Interventions: Procedure: Pain management

INTERVENTIONS:
Procedure: Pain management — Pain mamagement for burn care procedures.
  Other Names: Snow World or Standard of care
Other: Standard of care/no virtual reality game — no intervention for standard of care
  Other Names: Standard of care
  Arms: A

SUMMARY:
To examine the safety and efficacy of Virtual Reality (VR) distraction therapy in burn patients experiencing severe procedural pain during wound care.

DETAILED DESCRIPTION:
This is a prospective, randomized cross-over study of the safety and effectiveness of the use of a virtual reality distraction intervention to management procedural pain during burn wound care. Up to 20 subjects will be enrolled until 12 complete the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or oler with thermal injury
* Understands English
* patient perception of previous wound care procedural pain is greater than 6 on a numeric pain scal of 0-10 where 0= no pain and 10=worst pain ever experienced
* ability to use a computer mouse or hit the space bar on a computer keyboard

Exclusion Criteria:

* unhealed burned wounds on face, neck or head
* history of severe susceptibility to motion sickness
* presence of open woun ds to the hands that cannot be covered with a dressing while operating the control button
* patients who report a feeling of anxiety or discomfort while viewing the Snow World software on a computer without the helmet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
There will be a 20-50% reduction in pain while using Virtual Reality Games during burn wound care | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Maani, MD, Principal Investigator — United States Army Institute of Surgical Research
Locations (1):
- USAISR, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Patterson DR, Hoffman HG, Weichman SA, Jensen MP, Sharar SR. Optimizing control of pain from severe burns: a literature review. Am J Clin Hypn. 2004 Jul;47(1):43-54. doi: 10.1080/00029157.2004.10401474. No abstract available. PMID 15376608